CLINICAL TRIAL: NCT05549102
Title: The Impact of CBT on Shock-Potentiated Neural Circuity
Brief Title: CBT and the Neural Circuits of Anxiety
Status: Recruiting | Type: Observational
Sponsor: UCLH/UCL Joint Research Office (Other)
Collaborators: Medical Research Council (Other Government); Camden and Islington NHS Trust (Other Government); Central and North West London NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 121261; 255501 (Other: IRAS)
Record Dates: First submitted 2022-09-07; First posted 2022-09-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Generalised Anxiety Disorder; Anxiety Disorders; CBT; Anxiety Depression; Anxiety Disorders and Symptoms; Anxiety Generalized; Anxiety; Anxiety Disorder Generalized; Anxiety Disorder; Mixed With Depression (Mild)
Keywords: GAD; generalised anxiety disorder; anxiety disorders; cognitive behavioural therapy; CBT; psychological therapy; neural circuitry; emotional processing
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders; Lymphoma, Follicular | interventions — Cognitive Behavioral Therapy; Waiting Lists

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment Group: Participants undergoing a course of Cognitive Behavioural Therapy (CBT)
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Waiting List Group: Participants on the Waiting List for CBT
  Interventions: Other: Waiting List

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — In the Cognitive Behavioural Therapy group (N=87), patients will undergo CBT as part of their routine care in Step 3 of the IAPT programme. This will be administered by suitably trained clinicians. The specification of CBT is as recommended by the National Institute for Health and Care Excellence (NICE) guidelines (CG113 - Generalised anxiety disorder and panic disorder in adults: management). In these guidelines, patients are offered on average, 12-15 hourly, weekly sessions of CBT with a trained and competent practitioners. Therapy sessions involve discussions that identify patterns in thinking or behaviours which may be problematic, and therapists and patients work to set goals to reduce these using cognitive techniques. The principle is to teach the patient how to use CBT techniques in their day-to-day life to promote a lasting effect on mental health. We will test patients before (T1) and after (T2) a course of treatment.
  Other Names: CBT
  Groups: Treatment Group
Other: Waiting List — In the control group (N=87), we will test patients who are currently seeking (but not undergoing) treatment before (T1) and after a wait (T2) of equivalent time (i.e. waiting list controls)
  Groups: Waiting List Group

SUMMARY:
This study will aim to test whether specific neural circuitry changes, proposed on the basis of a neurocognitive model of anxiety, are a mechanism of action for Cognitive Behavioural Therapy (CBT) interventions. This study aims to provide a theoretical model of the neurobiological mechanisms of CBT's therapeutic effect, where there currently is none, and potentially allow for more targeted/specific approaches to anxiety disorders following the identification of key CBT mechanisms. The ultimate aim is to improve the efficacy of CBT, and more generally, psychological interventions for anxiety disorders.

DETAILED DESCRIPTION:
To test the hypothesis that the neural circuitry of the amygdala and prefrontal cortex will respond to CBT, the impact of a course of CBT on cortical-subcortical circuitry will be tested via a case-control study in individuals entering Improving Access to Psychological Therapies (IAPT) services (IAPT step 3; i.e., full CBT) for anxiety disorders and individuals in waiting lists. This design leverages the naturalistic waiting times in the clinical service and does not interfere with treatment as usual. Measures of brain region-specific connectivity and emotion-related behavioural performance will be assessed through testing sessions at the University College London (UCL) Institute of Cognitive Neuroscience and the Birkbeck-UCL Centre for NeuroImaging (BUCNI), involving computerised cognitive/psychological tasks and functional magnetic resonance imaging (fMRI).

The aims are to:

1. test whether this circuit responds to a course of CBT, by demonstrating disengagement of the circuit following CBT
2. relate this change in circuit function to behaviour through cognitive measures of emotional processing
3. explore the neurobiological features that distinguish patients who respond to CBT and those who do not
4. compare the data from this study to another on-going study assessing the impact of pharmacological interventions for anxiety, allowing for the comparison of neurobiological mechanisms of psychological vs. pharmacological treatments in anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in IAPT Step 3 (high intensity service)
* Score of or above 8 on the GAD-7 (indicating moderate anxiety on a standard scale of anxiety; Spitzer et al., 2006)
* Willing and able to provide written consent

Exclusion Criteria:

* Score above 22 on the GAD-7
* Past/present psychotic disorder, bipolar disorder/mania or alcohol/substance use disorder (outside a comorbid psychiatric episode)
* History of medical illness that may impair cognitive function (e.g. serious head injury, endocrine disorder)
* Current psychotropic pharmacological intervention (e.g. SSRIs) or use within 3 months
* MRI contraindications such as pacemaker, aneurysm clip, cochlear implant, neurostimulator, IUD, shrapnel, metal fragments in eye, weight of above 250lbs or claustrophobia
* Females who are pregnant, planning pregnancy, or breastfeeding

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Individuals entering IAPT services (IAPT step 3; i.e., full CBT) for anxiety disorders
Sampling Method: Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2020-02-02 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
'Aversive amplification circuit' connectivity | Day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  The engagement of the neural circuit of the amygdala, cingulate cortex and prefrontal cortex will be measured via an fMRI analysis technique called a psychophysiological interactions (PPI) analysis. PPI analysis concerns behaviour-specific increases in the relationship across regional brain activity - this means that it can allow one to assess whether two regions (a priori selected ROIs) show increased connectivity during a specific context or behaviour, suggesting a behaviour-specific increase in transfer of information. The output of this analysis will take form of a continuous beta weight - an index of connectivity across two brain regions (amygdala and medial prefrontal cortex), which represents the primary outcome of the study.

SECONDARY OUTCOMES:
Cognitive task performance: Loss/risk aversion task | Day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures how averse participants are to risk and loss in a mock gambling context
Cognitive task performance: Go/no-go task | Day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures approach/avoidance behaviours under threat of shock or safe conditions
Cognitive task performance: Facial emotional processing task | Day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures brain responses to positive, negative and neutral emotions
Cognitive task performance: Emotional face recognition task | Day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures brain responses during two distinct memory processes - the encoding (learning) and retrieval (remembering) of information
Cognitive task performance: Visual affective bias task | Day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures biases in patients' cognition towards or away from rewarding stimuli
Regional activations during neuroimaging task: Facial emotional processing task | Day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures brain responses to positive, negative and neutral emotions
Regional activations during neuroimaging task: Emotional face recognition task | Day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures brain responses during two distinct memory processes - the encoding (learning) and retrieval (remembering) of information
Regional activations during neuroimaging task: Visual affective bias task | Day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures biases in patients' cognition towards or away from rewarding stimuli
Clinical symptom measure: Generalised Anxiety Disorder Scale (GAD-7) | Screening, day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures symptoms of generalised anxiety, scored between 0-21 with higher scores indicating more severe symptoms
Clinical symptom measure: State Trait Anxiety Inventory (STAI) | Screening, day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures state and trait anxiety symptoms, scored between 20-80 with higher scores indicating more severe symptoms
Clinical symptom measures: Patient Health Questionnaire (PHQ-9) | Screening, day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures depressive symptoms, scored between 0-27 with higher scores indicating more severe symptoms
Clinical symptom measures: Beck's Depression Inventory (BDI) | Screening, day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures depressive symptoms, scored between 0-63 with higher scores indicating more severe symptoms
Clinical symptom measures: Catastrophizing questionnaire | Screening, day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures catastrophising, scored between 24-120 with higher scores indicating more severe symptoms
Clinical symptom measures: Daily Stress Inventory (DSI) | Screening, day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures frequency and impact of daily stresses. Frequency scored between 0-58 and impact scored between 0-6, with higher scores indicating more severe stress
Clinical symptom measures: Behavioural Inhibition/Behavioural Activation Scales (BIS/BAS) | Screening, day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures drive, fun-seeking, reward responsiveness and behavioural inhibition. Behavioural inhibition scored between 7-28, drive between 4-16, fun seeking between 4-16, and reward between 5-20, with higher scores indicating higher levels of those behaviours
Clinical symptom measures: Eysenck Impulsiveness Scale | Screening, day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  Measures impulsiveness, venturesomeness and empathy. Impulsivity scored between 0-19, venturesomeness between 0-16, empathy between 0-18, with higher scores indicating higher levels of those traits

OTHER OUTCOMES:
Mood diary | Day 0, up to 12 weeks (post-CBT or matched time on waiting list)
  A 'mood diary' will be implemented during the intervention phase which will involve daily self-report rating of mood ('happy', 'anxious' and 'sad')

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Cognitive Neuroscience, University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The data may also be published as open-access data online. In this case, all personally-identifiable data will be removed such that participants cannot be identified from this open data.